CLINICAL TRIAL: NCT01289418
Title: Short and Long-Term Electronic Surveillance of a Large Number of Healthcare Workers Following Administration of an Adjuvanted Ph1n1 Vaccine
Brief Title: Surveillance for Adverse Events Following Pandemic H1N1 Immunization
Status: Completed | Type: Observational
Sponsor: PHAC/CIHR Influenza Research Network (Other Government)
Collaborators: GlaxoSmithKline (Industry); Institut National en Santé Publique du Québec (Other); Laval University (Other); CHU de Quebec-Universite Laval (Other); Queen Elizabeth II Health Sciences Centre (Other); Mount Sinai Hospital, New York (Other); The Ottawa Hospital (Other); Hamilton Health Sciences Corporation (Other); Alberta Children's Hospital (Other); Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Gaston De Serres, Epidemiologist at the National Institute of Public Health of Quebec and professor of epidemiology at the University Laval, Laval University
Other Study IDs: pcirn-surveillancehcw-0910
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Novel Influenza A/H1N1
Keywords: H1N1; vaccine safety; adverse events; health care workers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Health care workers in Québec: Health care workers from CHUQ hospitals
- Health care workers in Toronto: Health care workers from the Mount Sinai Hospital
- Health care workers in Halifax: Health care workers from the Queen Elizabeth Hospital

SUMMARY:
Influenza vaccines are continuously modified to adjust to the virus antigenic shifts or drifts, and its safety profile may vary. While generally considered safe, influenza vaccines have been associated in the past with increases in cases of Guillain-Barré syndrome (1976) or with oculorespiratory syndrome (2001). The emergence of a novel strain of H1N1 influenza virus (pH1N1) has prompted health departments worldwide to prepare for mass vaccination campaigns with a new H1N1 pandemic vaccine. Following recommendations of the World Health Organization (WHO), Canada immunized its population with a dose-sparing adjuvanted vaccine. While the adjuvant developed by GlaxoSmithKline (GSK) has been administered to over 39 000 people, only a few hundred will have been vaccinated with the H1N1 formulation in clinical trials before the mass campaign was launched. With this small number, adverse events occurring at a rate < 1% will not be detected by these clinical trials.

Considering that most cases of pH1N1 to date have been relatively mild, it will be imperative to rapidly detect adverse events serious enough to reconsider the use of the vaccine. Passive surveillance is collecting notifications of adverse events but the sensitivity of this system is not high and its timeliness is not necessarily optimal.

In Canada, healthcare workers (HCW) are among those who were offered the new pandemic vaccine in priority. Because they were offered the vaccine early in the campaign and because they constitute a well-defined group in good general health, this group of people may be well suited for monitoring the safety of the pH1N1 vaccine.

The main objective of this project was to estimate in HCW vaccinated against pH1N1 the frequency of adverse events of sufficient severity to cause work absenteeism or medical consultation.

The active surveillance was done in HCW from 3 sites (Canadian hospitals) participating in the Pandemic Influenza Research Network (PCIRN): (1) Halifax (Nova Scotia), (2) Quebec City (Quebec): 3 hospitals, (3) Toronto

ELIGIBILITY:
Inclusion Criteria:

* To be a health care worker from one of the three Canadian Hospitals participating in the Public Health Agency of Canada/Canadian Institutes for Health Research- Influenza Research Network (PCIRN): Quebec City, Toronto, and Halifax.
* To have been immunized with the pH1N1 vaccine.
* To have an email address.
* To be 18 years old and older.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The active surveillance was conducted in three Canadian hospitals participating in the Public Health Agency of Canada/Canadian Institutes for Health Research- Influenza Research Network (PCIRN): Quebec City, Toronto, and Halifax. Healthcare workers immunized in these institutions were offered to participate in a web-based active surveillance of vaccine safety.
Sampling Method: Probability Sample
Enrollment: 6525 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaston De Serres, MD, PhD, Principal Investigator — Institut National en Santé Publique du Québec

REFERENCES:
- [Derived] De Serres G, Gariepy MC, Coleman B, Rouleau I, McNeil S, Benoit M, McGeer A, Ambrose A, Needham J, Bergeron C, Grenier C, Sleigh K, Kallos A, Ouakki M, Ouhoummane N, Stiver G, Valiquette L, McCarthy A, Bettinger J; PHAC-CIHR influenza Research Network (PCIRN). Short and long-term safety of the 2009 AS03-adjuvanted pandemic vaccine. PLoS One. 2012;7(7):e38563. doi: 10.1371/journal.pone.0038563. Epub 2012 Jul 3. PMID 22802929

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Care Workers: Health care workers from all hospitals
Period: Day 8 Survey
Arm/Group | Health Care Workers
Started | 6525
Completed | 4307
Not Completed | 2218
Not completed — email address invalid | 283
Not completed — participants did not complete the survey | 1935
Period: Day 29 Survey
Arm/Group | Health Care Workers
Started | 6525
Completed | 4057
Not Completed | 2468
Not completed — email address invalid | 283
Not completed — participants did not complete the survey | 2185

BASELINE CHARACTERISTICS:
Groups:
- Health Care Workers in Quebec: Health care workers from Quebec
- Health Care Workers in Toronto: Health Care Workers from Toronto
- Health Care Workers in Halifax: Health Care Workers from Halifax
- Total: Total of all reporting groups
Arm/Group | Health Care Workers in Quebec | Health Care Workers in Toronto | Health Care Workers in Halifax | Total
Number analyzed (Participants) | 5183 | 519 | 823 | 6525
Age Categorical [Number; unit: participants] — Demographic data was collected in only one site (n=3159). Some participants did not complete all the questions. That's why we don't have the age and the gender for all the participants.
  participants
    <=18 years | 0 | NA — demographic data were available only for Quebec | NA — demographic data were available only for Quebec | 0
    Between 18 and 65 years | 3152 | NA — demographic data were available only for Quebec | NA — demographic data were available only for Quebec | 3152
    >=65 years | 1 | NA — demographic data were available only for Quebec | NA — demographic data were available only for Quebec | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.7) | NA (NA) — demographic data were available only for Quebec | NA (NA) — demographic data were available only for Quebec | 37.5 (11.7)
Gender [Number; unit: participants] — Demographic data was collected in only one site (n=3159). Some participants did not complete all the questions. That's why we don't have the age and the gender for all the participants.
  participants
    Female | 2310 | NA — demographic data were available only for Quebec | NA — demographic data were available only for Quebec | 2310
    Male | 841 | NA — demographic data were available only for Quebec | NA — demographic data were available only for Quebec | 841
Region of Enrollment [Number; unit: participants]
  Canada | 5183 | 519 | 823 | 6525

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Experienced a New Health Problem or the Worsening of an Existing Health Condition That Resulted in a Medical Consultation.
Time Frame: at day 8, 15 and 29
Measure: Number; unit: participants
Groups:
- Health Care Workers: Health care workers with a valid e-mail address
Arm/Group | Health Care Workers
Number analyzed (Participants) | 6242
participants | 234

2. Primary Outcome: Number of Participants Who Had Experienced a New Health Problem or the Worsening of an Existing Health Condition That Resulted in Work Absenteeism.
Time Frame: day 8, 15 and 29
Measure: Number; unit: participants
Groups:
- Health Care Workers: Health care workers with a valid email address
Arm/Group | Health Care Workers
Number analyzed (Participants) | 6242
participants | 374

3. Primary Outcome: the Occurrence of Serious Adverse Events (SAE)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Health Care Workers From CHUQ Hospitals
Number analyzed (Participants) | 3064
participants | 35

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Health Care Workers From CHUQ Hospitals
Serious Adverse Events (participants affected / at risk) | 35/3064
Other Adverse Events (participants affected / at risk) | 383/4984
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Care Workers From CHUQ Hospitals (N=3064)
Breast cancer (Reproductive system and breast disorders) | 1 (1)
lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pancreas cancer (Endocrine disorders) | 1 (1)
cervix precancerous cells (Reproductive system and breast disorders) | 1 (1)
gynecologic problems/obstetrical (Pregnancy, puerperium and perinatal conditions) | 3 (3)
gynecologic problems (Reproductive system and breast disorders) | 3 (3)
Respiratory infection (Infections and infestations) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 4 (4)
cutaneous infection (Infections and infestations) | 2 (2)
toxic shock syndrome (Infections and infestations) | 1 (1)
abdominal problems (Gastrointestinal disorders) | 4 (4)
Musculoskeletal problems (Musculoskeletal and connective tissue disorders) | 2 (2)
depression (Psychiatric disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Chronic pericarditis (Cardiac disorders) | 1 (1)
Eye problem (Eye disorders) | 1 (1)
ear surgery (Surgical and medical procedures) | 1 (1)
severe headaches (General disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaso-vasectomy (Surgical and medical procedures) | 1 (1)
no diagnosis (Injury, poisoning and procedural complications) | 1 (1) — intermittent pain in the arm.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Care Workers From CHUQ Hospitals (N=4984)
Local reaction (Skin and subcutaneous tissue disorders) | 39 (39)
myalgia (General disorders) | 70 (70)
respiratory problems (Respiratory, thoracic and mediastinal disorders) | 201 (201)
gastroenteritis (Gastrointestinal disorders) | 73 (73)

LIMITATIONS AND CAVEATS:
Only 52% answered the 3 surveys. We don't know why 48% didn't complete the 3 surveys (were they too sick or not motivated).We didn't have a group of comparable unvaccinated individuals (to estimate the risks attributable to the vaccine).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No